CLINICAL TRIAL: NCT00934219
Title: Dose Related Decrease in Triglycerides in Patients With Hypertriglyceridemia and Treated With Lovaza.
Brief Title: Triglyceride Lowering Study
Acronym: TGLL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jewish Hospital, Cincinnati, Ohio (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Charles Glueck, MD Medical director of Cholesterol Center, Jewish Hospital Cholesterol Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TgLL8506
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-06

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia; triglycerides; familial hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type IV | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose Lovaza (Active Comparator): Lovaza 4 g twice a day, if not effective then 4 g 3 times a day
  Interventions: Drug: Omega-3-Acid Ethyl Esters
- Standard Dose (Active Comparator): 2 g twice a day
  Interventions: Drug: Omega-3-Acid Ethyl Esters

INTERVENTIONS:
Drug: Omega-3-Acid Ethyl Esters — LOVAZA, 1 g caps; High Dose Arm for 4 months, while on a standard therapy for hypertriglyceridemia (fibrates, +/-metformin). Standard Dose Arm for 3 months, while on a standard, unchanged therapy for hypertriglyceridemia (fibrates +/- metformin).
  Other Names: LOVAZA

SUMMARY:
Lovaza is a special fish oil concentrate, that prescribed at 4 g a day to reduce certain fat (triglycerides) levels in blood.Our goal is to study how Lovaza at doses of 4, 8, and 12 grams per day will reduce fats in the blood of the patients with very high level of triglycerides. Our hypothesis is that patients with very high triglycerides will respond more with higher doses of Lovaza (8 g per day and then 12 g per day).

DETAILED DESCRIPTION:
Lovaza contains Omega-3 fatty acids, the family of poly- unsaturated fatty acids. Omega-3 fatty acids stimulate blood circulation, increases the breakdown of fibrin, and additionally has been shown to reduce blood pressure, cardiac events and mortality from congestive heart failure. There is strong scientific evidence that omega 3 fatty acids significantly reduce blood triglyceride levels while elevating high density lipoprotein cholesterol (HDL) levels. Fasting and non fasting hypertriglyceridemia have been associated with atherosclerosis, and coronary heart disease events, even in the absence of hypercholesterolemia. Severe hypertriglyceridemia (>2000 mg/dl) can also lead to acute hemorrhagic pancreatitis.

Currently, patients having very High TG are treated with Fibric acids (gemfibrozil, Tricor, Antara), and if hyperinsulinemic, with Glucophage. Lovaza (4g/day) has been shown to be effective and safe in lowering TG levels. There is no published data which indicates that Lovaza 8 or 12 g per day would have therapeutic effectiveness in further normalizing triglycerides in subjects on maximized triglyceride lowering and Lovaza 4 g per day. We hypothesize, based on our clinical experience that increasing Lovaza to 8 and then (if necessary) to 12 g/day would safely optimize triglycerides in subjects with primary hypertriglyceridemia who failed to normalize their triglycerides on optimal therapy including Lovaza 4 g/day.

ELIGIBILITY:
Inclusion Criteria:

1. Primary hypertriglyceridemia with fasting TG levels >1000 mg/dl, and persistence of TG levels > 500 mg/dl despite maximal TG lowering therapy for 1 month, including Lovaza 4 g/day, fibric acids, and, where indicated, Glucophage for treatment of hyperinsulinemia.
2. Patients with mild to moderately impaired renal function should be initiated on TRICOR 48 mg and patients with severe renal impairment should not be given TRICOR.
3. Absence of exclusionary criteria (see below).

Exclusion Criteria:

1. Patients with known allergy to fish
2. Hypertriglyceridemia secondary to alcoholism, exogenous estrogens, nephrotic syndrome, hemochromatosis, glycogen storage disease, uncontrolled diabetes, exogenous corticosteroids, Cushing's syndrome, uremia).
3. Bleeding gastric or duodenal ulcers, active inflammatory bowel disease.
4. Pregnancy
5. Dementia
6. Patients with bleeding diatheses
7. Patients who are taking concomitant anticoagulants and other medications that affect bleeding time (e.g., warfarin, aspirin)
8. Patients with significantly abnormal transaminases (above 3x of upper normal limit)or any history of liver disease
9. Patients with conditions affecting the skin (e.g. malignancy, vasculitides) that may confound the skin exam.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
triglycerides level | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Glueck, MD, Principal Investigator — JEWISH HOSPITAL CHOLESTEROL CENTER
Locations (1):
- Jewish Hospital Cholesterol Center, Cincinnati, Ohio, United States

REFERENCES:
- See also: Free Triglycerides lowering study — http://www.jewishhospitalcincinnati.com/cholesterol/Research/FREE_TRIGLYCERIDE_LOWERING_STUDY-2009.html